CLINICAL TRIAL: NCT04314453
Title: Comparisons of TESSYS and "U" Route Procedures of Transforaminal Percutaneous Endoscopic Lumbar Discectomy on Lumbar Spinal Stenosis Treatment
Brief Title: Comparisons Therapeutic Effects of Different PELD Procedure on LSS.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, BINBIN WU, Attending Doctor, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2020-14-206
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Degeneration Disc; Lumbar Spinal Stenosis
Keywords: percutaneous endoscopic lumbar discectomy; minimally invasive; transforaminal endoscopic spine system; U route
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T group: The degenerative lumbar spinal stenosis patients accepted the PELD with TESSYS procedure.
  Interventions: Other: percutaneous endoscopic lumbar discectomy
- U group: The degenerative lumbar spinal stenosis patients accepted the PELD with U route procedure.
  Interventions: Other: percutaneous endoscopic lumbar discectomy

INTERVENTIONS:
Other: percutaneous endoscopic lumbar discectomy — Resection of the hypertrophied faceted joints, osteophyte formation and ligamentum flavum (LF) hypertrophy, with or without disc protrusion for degenerative spinal stenosis.

SUMMARY:
Different procedure of percutaneous endoscopic lumbar discectomy (PELD) was with ventral decompression of dural sac on the lumbar spinal stenosis remains unkonwn.The traditional transforaminal endoscopic spine system (TESSYS) of PELD has been used in clnical for many years, but cannot achieve dorsal decompression. A newly developed modified TESSYS procedure, "U" route PELD combining ventral and dorsal decompression was introduced. Nevertheless, the superior between TESSYS and "U" route PELD procedures on treating LSS remains unknown. This study is desinged to recruit degenerative lumbar spinal stenosis patients who underwent TESSYS or "U" rout PELD, recruited from January 2014 to December 2017. These patients will be followed up for 2 years, and assessed the minimum dura sac cross sectional area (mDCSA) by MRI, and visual analogue scale (VAS) and Oswestry Disability Index (ODI) at pre- and post-operation. The global clinical outcomes were evaluated using modified MacNab criteria postoperatively. Thus, comprehensively evaluate the safety and therapeutic effects of the two PELD procedures on LSS treatments.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with the diagnosis of degenerative lumbar spinal stenosis (LSS) (central stenosis with or without lateral recess stenosis) on mono or double segments, with the imaging evidence of magnetic resonance images (MRI) and computed tomography (CT); (2) patients presented low back pain, limp and sciatica, and have accepted conservative treatment more than 3 months but failed in symptoms relief; (3) patients agreed to accept TESSYS or the "U" route PELD procedure over other spinal surgeries; (4) patients had lumbar MRI imaging examines in our hospital at pre- and post-operation.

Exclusion Criteria:

* (1) patients with spinal instability, including dynamic instability or more than Grade II spondylolisthesis; (2) patients had spinal surgical history; (3) patients with peripheral nerve disease, systematic infection, bleeding diathesis or high risk of bleeding that cannot tolerate the surgery; (4) patients with mental illness and were uncooperative; (5) patients lost to the follow up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The degenerative lumbar spinal stenosis patients who underwent TESSYS or "U" rout PELD, recruited from January 2014 to December 2017.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Pain assessed by Visual Analogue Scale | Preoperation to postoperative 2 years.
  Visual Analogue Scale (VAS 0 to 10)
Oswestry Disability Index (ODI) | Preoperation to postoperative 2 years.
  the disability with ODI (0 to 100)

SECONDARY OUTCOMES:
minimum Dural sac cross sectional area (mDCSA) | Baseline and postoperative 1-month
  the mDCSA at the most constricted lumbar spinal level of surgical intervertebral disc were measured for three times by the software of INFINITT Picture Archiving and Communication System (PACS) (INFINITT Healthcare Co., Seoul Korea)

IPD SHARING:
Plan to Share IPD: No